CLINICAL TRIAL: NCT03592615
Title: Prevalence of Binocular Vision Anomalies Before and After Cataract and Refractive Surgery
Brief Title: Binocular Vision Anomalies After Cataract and Refractive Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Salus University (Other)
Responsible Party: Principal Investigator, Qing-Qing Tan, PhD student, Salus University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: qqt0001
Record Dates: First submitted 2018-06-08; First posted 2018-07-19 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Binocular Vision Disorder; Refractive Errors; Cataract
Keywords: prevalence; binocular vision disorders; accommodative disorders; cataract surgery; corneal refractive surgery
MeSH Terms: conditions — Refractive Errors; Cataract | interventions — Cataract Extraction; Phacoemulsification; Keratomileusis, Laser In Situ; Keratectomy, Subepithelial, Laser-Assisted

STUDY DESIGN:
Intervention Model Description: Cataract group: participants undergo cataract surgery for vision correction Refractive error group: participants undergo corneal refractive surgery for vision correction
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cataract group (Experimental): All participants in this arm undergo cataract surgery for the purpose of vision correction.
  Interventions: Procedure: cataract surgery
- Refractive error group (Experimental): All participants in this arm undergo corneal refractive surgery for the purpose of vision correction.
  Interventions: Procedure: Corneal refractive surgery

INTERVENTIONS:
Procedure: cataract surgery — Cataract surgery in this study is only for the purpose of vision correction, not for the treatment of ocular pathology other than cataract, e.g., treatment for lens dislocation. The surgery used in this study should not be combined with other procedures, such as limbal relaxing incision for treating astigmatism.
  Other Names: phacoemulsification; cataract extraction
  Arms: Cataract group
Procedure: Corneal refractive surgery — Corneal refractive surgery in this study is only for the purpose of vision correction, not for the treatment of ocular pathology other than refractive error, e.g., treatment for corneal scar. The surgery used in this study should not be combined with other procedures, such as limbal relaxing incision for treating severe astigmatism.
  Other Names: LASIK; LASEK; PRK; SMILE
  Arms: Refractive error group

SUMMARY:
There are indications in the literature that binocular vision disorders may occur after cataract and corneal refractive surgery. It is not clear whether these problems are new or represent decompensation of previously existing conditions. However, the following significant study limitations exist in the current literature: 1) lack of attention to non-strabismic binocular vision disorders, 2) incomplete binocular vision assessment, 3) a validated symptom survey was not used, 4) diplopia was typically the only symptom studied, 5) retrospective study design, and 6) in the few prospective studies the sample sizes were small.

Given the limitations in the current literature there is a need for further study of the prevalence and significance of binocular vision problems after cataract surgery and binocular vision and accommodative problems after corneal refractive surgery.

This study aims to determine whether there is an increase in the prevalence of binocular vision problems after cataract surgery and accommodative and binocular vision disorders after refractive surgery.

DETAILED DESCRIPTION:
1. Research plan Specific aim 1A: To investigate the prevalence of non-strabismic and strabismic binocular vision anomalies after cataract surgery. Specific aim 1B: To investigate the prevalence accommodative and binocular vision disorders after refractive surgery. Specific aim 2: To determine if increase in the prevalence of binocular anomalies is different for cataract surgery compared to refractive surgery. Specific aim 3: To develop an efficient examination protocol that would enable eye care professionals to determine if a patient is at risk for binocular vision anomalies after cataract surgery and accommodative and binocular vision disorders after refractive surgery.

   The proposed study will address the weaknesses in the current literature. The study will be prospective and will use explicit and well-defined eligibility and exclusion criteria. A comprehensive battery of accommodative (pre-presbyopes only) and binocular vision tests will be administered on all the patients before the surgery of the first eye and 12 weeks after the surgery of the second eye.

   A pre-defined classification protocol will be used to determine if a binocular vision disorder is present before surgery, after surgery, or whether there has been a change in the condition after surgery.

   A total prevalence of postoperative strabismic and non-strabismic binocular vision anomalies will be determined for the cataract population and the refractive error group.
2. Statistical analysis plan 2.1 Specific aim 1A Hypothesis: There will be a statistically significant increase in the prevalence of binocular vision anomalies after cataract surgery

A sample size calculation based on a McNemar's test to compare the prevalence of binocular vision anomalies before and after cataract surgery was performed using the Power and Sample Size Program (PS version 3.1.2). Base on a previous literature, the overall prevalence of accommodative and binocular vision anomalies in adult population (18-35 years) is 13.15%. However, no existing literature reported the prevalence of binocular vision anomalies after cataract surgery.

We propose that 15% increase in prevalence is clinically meaningful. The correlation between paired observations is 0.2, as recommended by Dupont. Although this is a large effect, the effect of cataract surgery on prevalence of binocular vision anomalies may be this large (presumed by an experienced binocular vision specialist). If the effect is smaller and the difference not statistically significant, the study will provide valuable data to plan another study. Therefore, a sample size calculation suggests that a total of 44 participants will yield a power of 80% with a significant level of 5%. To account for potential loss to follow-up, a sample size of 50 will be selected for the cataract group. All analyses will be performed using SPSS Statistics 24.0 with an alpha level of 0.05 to determine the statistical significance. A calculation for the prevalence of binocular vision anomalies before and after surgery will be performed. A two-tailed McNemar's Chi-Square Test will be used to test the statistical significance of the change in the proportion of binocular vision anomalies before and after surgery.

2.2 Specific aim 1B Hypothesis: There will be a statistically significant increase in the prevalence of binocular vision and accommodative anomalies after refractive surgery.

The sample size calculation process for specific aim 1B was the same as for specific aim 1A. Therefore, a sample size of 50 will also be selected for the refractive error group. A calculation for the prevalence of accommodative and binocular vision anomalies before and after surgery will be performed. A two-tailed McNemar's Chi-Square Test will be used to test the statistical significance of the changes in the proportions of binocular vision anomalies before and after surgery.

2.3 Specific aim 2 Hypothesis: The increase in prevalence of binocular vision anomalies will be greater after cataract surgery than refractive surgery.

A calculation for the prevalence of binocular vision anomalies will be performed respectively in the cataract group and the refractive error group. A two-tailed Contingency Chi-Square Test will be used to test the statistical significance of difference of changes in the proportion of binocular vision anomalies before and after surgery in both groups.

2.4 Specific aim 3 Hypothesis: A short screening protocol will be of equal effectiveness to a comprehensive assessment of binocular vision and accommodation to determine which patients may be at risk for post-surgical binocular vision and accommodative anomalies.

A two-tailed MacNemar's Chi-Square Test will be used to test the statistical significance of difference in the effectiveness of a short screening protocol and a comprehensive assessment for determining the risk for post-surgical binocular vision and accommodative anomalies. Sensitivity and specificity for the short screening protocol will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Cataract patients who are willing to undergo cataract extraction and intraocular lens implantation
* Refractive error patients who are willing to undergo laser corneal refractive surgery
* 18 years and older in cataract group
* 18-35 years old in refractive error group
* Any gender
* Any race or ethnicity
* Informed consent and willingness to participate in the study

Exclusion Criteria:

* Other ocular pathology that affect vision and binocular alignment in addition to cataract or refractive error
* Surgical complications that may affect binocular vision testing, such as a subluxation of the IOLs or macular edema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Changes from pre-surgical phoria at 12 weeks post surgery | Pre-surgery and 12 weeks post surgery
  Phoria will be measured using cover test (in prism diopters).
Changes from pre-surgical fusional vergence at 12 weeks post surgery | Pre-surgery and 12 weeks post surgery
  Fusional vergence will be measured using step vergence testing (in prism diopters).
Changes from pre-surgical convergence amplitude at 12 weeks post surgery | Pre-surgery and 12 weeks post surgery
  Convergence amplitude will be measured using near point of convergence test (in centimeters).
Changes from pre-surgical vergence facility at 12 weeks post surgery | Pre-surgery and 12 weeks post surgery
  Vergence facility will be measured using vergence facility testing (in cycle per minute).
Changes from pre-surgical accommodative amplitude at 12 weeks post surgery (refractive error group only) | Pre-surgery and 12 weeks post surgery
  Accommodative amplitude will be measured using monocular amplitude of accommodation testing (in diopters).
Changes from pre-surgical accommodative facility at 12 weeks post surgery (refractive error group only) | Pre-surgery and 12 weeks post surgery
  Accommodative facility will be measured using monocular accommodative facility testing (in cycle per minute).

SECONDARY OUTCOMES:
changes from pre-surgical stereopsis at 12 weeks post surgery | pre-surgery and 12 weeks post surgery
  Randot stereo test (recorded in second of arc)
changes from pre-surgical aniseikonia at 12 weeks post surgery | pre-surgery and 12 weeks post surgery
  Aniseikonia Inspector Software Program (recorded in percentage)
changes from pre-surgical CISS score at 12 weeks post surgery | pre-surgery and 12 weeks post surgery
  Convergence insufficiency symptom survey (recorded in a summation of the CISS score). The CISS is a 15-items survey questioning the participants whether they have the symptoms related to binocular vision disorders. Each item has a scale ranging from 0 to 4, of which 0=never, 1=not very often, 2=sometimes, 3=fairly often, 4=always. A higher score indicates a worse outcome. The total score will be summed from the 15 items.

CONTACTS AND LOCATIONS:
Overall Officials: Qing-Qing Tan, MSc, Principal Investigator — Salus University
Locations (1):
- Salus University, Elkins Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Minnal VR, Rosenberg JB. Refractive surgery: a treatment for and a cause of strabismus. Curr Opin Ophthalmol. 2011 Jul;22(4):222-5. doi: 10.1097/ICU.0b013e3283477c60. PMID 21537187
- [Background] Kalantzis G, Papaconstantinou D, Karagiannis D, Koutsandrea C, Stavropoulou D, Georgalas I. Post-cataract surgery diplopia: aetiology, management and prevention. Clin Exp Optom. 2014 Sep;97(5):407-10. doi: 10.1111/cxo.12197. PMID 25138745
- [Background] Gawecki M, Grzybowski A. Diplopia as the Complication of Cataract Surgery. J Ophthalmol. 2016;2016:2728712. doi: 10.1155/2016/2728712. Epub 2016 Feb 21. PMID 26998351
- [Background] Finlay AL. Binocular vision and refractive surgery. Cont Lens Anterior Eye. 2007 May;30(2):76-83. doi: 10.1016/j.clae.2007.02.009. PMID 17448926
- [Background] Loba P, Rajska K, Simiera J, Wilczynski M, Omulecki W, Broniarczyk-Loba A. The influence of a prolonged interoperative period on binocular vision after bilateral cataract extractions. Eur J Ophthalmol. 2015 Jul-Aug;25(4):315-9. doi: 10.5301/ejo.5000569. Epub 2015 Jan 27. PMID 25633621
- [Background] Rutstein RP, Fullard RJ, Wilson JA, Gordon A. Aniseikonia induced by cataract surgery and its effect on binocular vision. Optom Vis Sci. 2015 Feb;92(2):201-7. doi: 10.1097/OPX.0000000000000491. PMID 25546829
- [Background] Chung SA, Kim CY, Chang JH, Hong S, Kang SY, Seong GJ, Lee JB. Change in ocular alignment after topical anesthetic cataract surgery. Graefes Arch Clin Exp Ophthalmol. 2009 Sep;247(9):1269-72. doi: 10.1007/s00417-009-1084-8. Epub 2009 Apr 30. PMID 19404663
- [Background] Golnik KC, West CE, Kaye E, Corcoran KT, Cionni RJ. Incidence of ocular misalignment and diplopia after uneventful cataract surgery. J Cataract Refract Surg. 2000 Aug;26(8):1205-9. doi: 10.1016/s0886-3350(00)00330-8. PMID 11008049
- [Background] Nayak H, Kersey JP, Oystreck DT, Cline RA, Lyons CJ. Diplopia following cataract surgery: a review of 150 patients. Eye (Lond). 2008 Aug;22(8):1057-64. doi: 10.1038/sj.eye.6702847. Epub 2007 Apr 27. PMID 17464297
- [Background] Karagiannis D, Chatzistefanou K, Damanakis A. Prevalence of diplopia related to cataract surgery among cases of diplopia. Eur J Ophthalmol. 2007 Nov-Dec;17(6):914-8. doi: 10.1177/112067210701700608. PMID 18050117
- [Background] Hutchinson AK. Refractive surgery for accommodative esotropia: past, present, and future. Eur J Ophthalmol. 2012 Nov-Dec;22(6):871-7. doi: 10.5301/ejo.5000210. Epub 2012 Oct 10. PMID 23097019
- [Background] Kirwan C, O'Keefe M, O'Mullane GM, Sheehan C. Refractive surgery in patients with accommodative and non-accommodative strabismus: 1-year prospective follow-up. Br J Ophthalmol. 2010 Jul;94(7):898-902. doi: 10.1136/bjo.2009.162420. Epub 2009 Nov 30. PMID 19948562
- [Background] Snir M, Kremer I, Weinberger D, Sherf I, Axer-Siegel R. Decompensation of exodeviation after corneal refractive surgery for moderate to high myopia. Ophthalmic Surg Lasers Imaging. 2003 Sep-Oct;34(5):363-70. PMID 14509458
- [Background] Kushner BJ, Kowal L. Diplopia after refractive surgery: occurrence and prevention. Arch Ophthalmol. 2003 Mar;121(3):315-21. doi: 10.1001/archopht.121.3.315. PMID 12617699
- [Background] Chung SA, Kim WK, Moon JW, Yang H, Kim JK, Lee SB, Lee JB. Impact of laser refractive surgery on ocular alignment in myopic patients. Eye (Lond). 2014 Nov;28(11):1321-7. doi: 10.1038/eye.2014.209. Epub 2014 Sep 5. PMID 25190533
- [Background] Prakash G, Choudhary V, Sharma N, Titiyal JS. Change in the accommodative convergence per unit of accommodation ratio after bilateral laser in situ keratomileusis for myopia in orthotropic patients: prospective evaluation. J Cataract Refract Surg. 2007 Dec;33(12):2054-6. doi: 10.1016/j.jcrs.2007.07.030. PMID 18053903
- [Background] Han J, Hong S, Lee S, Kim JK, Lee HK, Han SH. Changes in fusional vergence amplitudes after laser refractive surgery for moderate myopia. J Cataract Refract Surg. 2014 Oct;40(10):1670-5. doi: 10.1016/j.jcrs.2014.01.043. Epub 2014 Aug 20. PMID 25149555
- [Background] Li M, Cheng H, Yuan Y, Wang J, Chen Q, Me R, Ke B. Change in choroidal thickness and the relationship with accommodation following myopic excimer laser surgery. Eye (Lond). 2016 Jul;30(7):972-8. doi: 10.1038/eye.2016.75. Epub 2016 Apr 15. PMID 27080489
- [Background] Zheng K, Han T, Zhou X. Accommodative changes after SMILE for moderate to high myopia correction. BMC Ophthalmol. 2016 Oct 4;16(1):173. doi: 10.1186/s12886-016-0352-8. PMID 27716112
- [Background] Karimian F, Baradaran-Rafii A, Bagheri A, Eslani M, Bayat H, Aramesh S, Yaseri M, Amin-Shokravi A. Accommodative changes after photorefractive keratectomy in myopic eyes. Optom Vis Sci. 2010 Nov;87(11):833-8. doi: 10.1097/OPX.0b013e3181f6fccc. PMID 20871473
- [Background] Wylie J, Henderson M, Doyle M, Hickey-Dwyer M. Persistent binocular diplopia following cataract surgery: aetiology and management. Eye (Lond). 1994;8 ( Pt 5):543-6. doi: 10.1038/eye.1994.134. PMID 7835450
- [Background] Godts D, Trau R, Tassignon MJ. Effect of refractive surgery on binocular vision and ocular alignment in patients with manifest or intermittent strabismus. Br J Ophthalmol. 2006 Nov;90(11):1410-3. doi: 10.1136/bjo.2006.090902. Epub 2006 Aug 2. PMID 16885192
- [Background] Brugnoli de Pagano OM, Pagano GL. Laser in situ keratomileusis for the treatment of refractive accommodative esotropia. Ophthalmology. 2012 Jan;119(1):159-63. doi: 10.1016/j.ophtha.2011.07.003. Epub 2011 Sep 29. PMID 21959372
- [Background] Giannaccare G, Primavera L, Fresina M. Photorefractive keratectomy influences the angle of ocular deviation in strabismus patients with hyperopia. Int Ophthalmol. 2019 Apr;39(4):737-744. doi: 10.1007/s10792-018-0867-5. Epub 2018 Mar 3. PMID 29502213
- [Background] Garcia-Munoz A, Carbonell-Bonete S, Canto-Cerdan M, Cacho-Martinez P. Accommodative and binocular dysfunctions: prevalence in a randomised sample of university students. Clin Exp Optom. 2016 Jul;99(4):313-21. doi: 10.1111/cxo.12376. Epub 2016 Mar 29. PMID 27027297
- [Background] Dupont WD. Power calculations for matched case-control studies. Biometrics. 1988 Dec;44(4):1157-68. PMID 3233252
- [Derived] Tan QQ, Tan JH, Luo CK, Lai CY, Zhao W, Lan CJ, Lewis J, Aljohani S, Liao X, Scheiman M. A brief effective screening protocol for identifying cataract patients with binocular vision anomalies. BMC Ophthalmol. 2024 Dec 18;24(1):536. doi: 10.1186/s12886-024-03807-w. PMID 39695508
- [Derived] Tan QQ, Lewis JS, Lan CJ, Liao X, Tang XL, Wang J, Aljohani S, Scheiman MM. Cataract surgery is not associated with post-operative binocular vision anomalies in age-related cataract patients. Ophthalmic Physiol Opt. 2022 Sep;42(5):998-1008. doi: 10.1111/opo.13012. Epub 2022 Jun 12. PMID 35690924
- [Derived] Tan QQ, Lewis JS, Lan CJ, Liao X, Tang XL, Wang J, Scheiman MM. Preoperative binocular vision characteristics in the age-related cataract population. BMC Ophthalmol. 2022 Apr 27;22(1):196. doi: 10.1186/s12886-022-02418-7. PMID 35477368